CLINICAL TRIAL: NCT01020019
Title: A Randomized, Double-Blind, Placebo-Controlled Study of Lofexidine and Dronabinol for the Treatment of Marijuana Dependence
Brief Title: Combined Pharmacotherapy for Cannabis Dependency
Acronym: D-LUCS
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Frances R Levin, Director of Substance Use Disorder, National Institute on Drug Abuse (NIDA)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: #6015; P50DA009236-16 (NIH)
Record Dates: First submitted 2009-11-24; First posted 2009-11-25 (Estimated); Results first posted 2016-05-11 (Estimated); Last update posted 2019-04-24 (Actual); Status verified 2019-04

CONDITIONS: Cannabis Dependence; Marijuana Dependence
Keywords: Cannabis Dependence; Marijuana Dependence; Marinol; Lofexidine
MeSH Terms: conditions — Marijuana Abuse | interventions — Dronabinol; lofexidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lofexidine and Dronabinol (Experimental): Maintained at 1.8mg/day Lofex. and 60 mg/day of Dronabinol
  Interventions: Drug: Dronabinol; Drug: Lofexidine
- Placebo (Placebo Comparator): Lofex. matched placebo Dronabinol placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dronabinol — Dronabinol: 20 mg/TID
  Other Names: Marinol
  Arms: Lofexidine and Dronabinol
Drug: Placebo — Placebo control
  Arms: Placebo
Drug: Lofexidine — Lofex: .6 mg/ TID
  Arms: Lofexidine and Dronabinol

SUMMARY:
The purpose of this study is to see if Lofexidine in combination with Marinol is superior to placebo in achieving abstinence, reducing cannabis use and reducing withdrawal in cannabis-dependent patients seeking treatment for their marijuana use.

DETAILED DESCRIPTION:
Cannabis use disorders remain the most common illicit drug use disorder and options for treatment remain limited. Compared to other abusable substances, there has been little investigation of pharmacotherapies for cannabis dependence and no effective pharmacotherapy for cannabis dependence has yet to been developed. The development of effective cannabis dependence pharmacotherapy is an important unmet public health need. Agonist pharmacotherapy strategies have been effective for other substance use disorders (e.g., opioid and nicotine use disorders) and the endocannabinoid system represents a promising target for agonist pharmacotherapy with dronabinol. Lofexidine, a noradrenergic system suppressant, is effective in treating opioid withdrawal and shows promise as a cannabis use disorder pharmacotherapy. Haney et al. (2008) found that the combination of lofexidine and dronabinol (Lofex-Dro) was superior to placebo, lofexidine alone, or dronabinol alone in improving sleep and other cannabis withdrawal symptoms. Further, reduction in craving and relapse was greater for this combined pharmacotherapy relative to either medication alone or placebo. The proposed protocol is a 2 group, double blind, placebo-controlled outpatient study of the safety and efficacy of the combination of dronabinol and lofexidine for the treatment of cannabis dependence. We plan to enroll 180 subjects in a 12-week trial. The primary hypothesis is that dronabinol will act as an agonist treatment while lofexidine will suppress craving- and cue-induced related stress such that the combination will act in a complementary manner to induce prolonged abstinence from marijuana.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women between the ages of 18-60 who meet DSM-IV criteria for current marijuana dependence
2. Individuals must report using marijuana at least 5 days a week and have a positive urine test for THC on the day of study entry.
3. Individual must describe marijuana as their primary drug of abuse.
4. Individuals must be capable of giving informed consent and capable of complying with study procedures.

Exclusion Criteria:

1. Meets DSM-IV-TR criteria for schizophrenia, schizoaffective illness, psychotic disorder other than transient psychosis due to drug abuse, major depression, bipolar illness or psychiatric disorders (other than substance abuse) which require psychiatric intervention.
2. Individuals who are medically unstable based on laboratory tests, electrocardiogram, medical history, physical examination that would make participation hazardous
3. Individuals with liver enzyme function tests greater than three times normal
4. Individuals with a history of seizure disorder
5. Individuals with current suicidal risk.
6. Individuals who are cognitively impaired
7. Bradycardia (< 50 beats/minute), hypotension (sitting or standing BP < 90/50), or symptoms attributable to low BP (i.e. lightheadedness or dizziness on standing).
8. Nursing mothers and pregnant women. Women of child bearing age will be included in the study provided that they are not pregnant, based on the results of a blood pregnancy test drawn at the time of screening. They must also agree to use a method of contraception with proven efficacy and agree not to become pregnant during the study. To confirm this, urine pregnancy tests will be repeated monthly. Women will be provided a full explanation of the potential dangers of pregnancy while on the study medication. If a woman becomes pregnant, the study medication will be discontinued.
9. Individuals who are physiologically dependent on any other drugs (excluding nicotine) that would require a medical intervention
10. Individuals with known sensitivity to dronabinol or lofexidine
11. Individuals with coronary vascular disease as indicated by history or suspected by abnormal ECG or history of cardiac symptoms
12. Individuals currently being treated with an alpha-2 agonist antihypertensive medication
13. Individuals currently being prescribed a psychotropic medication (including sleep medication). However, medication for depression is allowed if stable for at least 1 month.
14. Individuals who have a job that even mild intoxication would be hazardous (e.g., firefighter, bus driver)
15. Individuals who are court-mandated to treatment.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 156 (Actual)
Dates: Start 2010-01; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Frances R Levin, M.D., Principal Investigator — Columbia University
Locations (1):
- New York State Psychiatric Institute, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Brezing CA, Choi CJ, Pavlicova M, Brooks D, Mahony AL, Mariani JJ, Levin FR. Abstinence and reduced frequency of use are associated with improvements in quality of life among treatment-seekers with cannabis use disorder. Am J Addict. 2018 Mar;27(2):101-107. doi: 10.1111/ajad.12660. Epub 2018 Feb 19. PMID 29457671

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were treated at the Substance Treatment and Research Service (STARS) of Columbia University/ New York State Psychiatric Institute (NYSPI). Study enrollment occurred from January 2010 through May 2014 with study completion in September 2014.
Pre-assignment Details: The study included a one-week placebo lead-in phase. Participants were randomized at the end of the placebo lead-in phase and those who reported marijuana use less than once a week during the lead-in phase were considered placebo responders and were not randomized. A total of 34 participants discontinued prior to randomization for various reasons.
Groups:
- Lofexidine and Dronabinol: Maintained at 1.8mg/day Lofex. and 60 mg/day of Dronabinol
  Lofexidine and Dronabinol: Lofex: .6 mg/ TID Dronabinol: 20 mg/TID
Period: Overall Study
Arm/Group | Placebo | Lofexidine and Dronabinol
Started | 61 | 61
Completed | 35 | 32
Not Completed | 26 | 29
Not completed — Lost to Follow-up | 21 | 18
Not completed — Adverse Event | 1 | 5
Not completed — not interested in treatment | 4 | 4
Not completed — moving | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Lofexidine and Dronabinol | Total
Number analyzed (Participants) | 61 | 61 | 122
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.4 (10.8) | 34.8 (11.2) | 35.2 (10.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 22 | 38
  Male | 45 | 39 | 84
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic | 15 | 17 | 32
  Black | 17 | 18 | 35
  White | 26 | 21 | 47
  Other | 3 | 5 | 8

OUTCOME MEASURES:

1. Primary Outcome: 21 Days of Consecutive Abstinence as Measured by the Time-line Followback.
Time Frame: reported daily for 12 weeks/ or study participation
Measure: Number; unit: participants
Arm/Group | Placebo | Lofexidine and Dronabinol
Number analyzed (Participants) | 61 | 61
participants | 18 | 17

ADVERSE EVENTS:
Time Frame: 12 weeks of trial or participants length of participation
Arm/Group | Placebo | Lofexidine and Dronabinol
Serious Adverse Events (participants affected / at risk) | 1/61 | 1/61
Other Adverse Events (participants affected / at risk) | 46/61 | 47/61
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=61) | Lofexidine and Dronabinol (N=61)
abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
detoxification (Psychiatric disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=61) | Lofexidine and Dronabinol (N=61)
dry mouth (General disorders) | 6 (6) | 27 (27)
fatigue (General disorders) | 15 (15) | 26 (26)
dizzy (General disorders) | 12 (12) | 21 (21)
insomnia (General disorders) | 13 (13) | 13 (13)
intoxication (General disorders) | 2 (2) | 13 (13)
headache (General disorders) | 12 (12) | 10 (10)
anxiety (Psychiatric disorders) | 11 (11) | 3 (3)
hypotension (Vascular disorders) | 1 (1) | 10 (10)
drowsiness (General disorders) | 4 (4) | 9 (9)
upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 8 (8) | 2 (2)
nausea (Gastrointestinal disorders) | 5 (5) | 6 (6)
irritability (General disorders) | 6 (6) | 3 (3)
decreased appetite (Metabolism and nutrition disorders) | 6 (6) | 2 (2)
sweating (Skin and subcutaneous tissue disorders) | 5 (5) | 5 (5)
depression (Psychiatric disorders) | 5 (5) | 3 (3)
stomache upset (Gastrointestinal disorders) | 5 (5) | 2 (2)
diarrhea (Gastrointestinal disorders) | 4 (4) | 2 (2)
vomitting (Gastrointestinal disorders) | 4 (4) | 2 (2)
fever (General disorders) | 4 (4) | 1 (1)
orthostasis (Vascular disorders) | 1 (1) | 4 (4)
sore throat (General disorders) | 3 (3) | 2 (2)
gas (Gastrointestinal disorders) | 1 (1) | 3 (3)
confusion (Nervous system disorders) | 1 (1) | 3 (3)
rash (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No